CLINICAL TRIAL: NCT03606330
Title: Systemic, Pancoronary and Local Plaque Vulnerability for Image-based Prediction of Acute Coronary Syndromes - the VIP Study
Brief Title: Systemic, Pancoronary and Local Coronary Vulnerability
Acronym: VIP
Status: Completed | Type: Observational
Sponsor: Cardio Med Medical Center (Industry)
Collaborators: University of Targu Mures, Romania (Other); University Hospital of Targu Mures, Romania (Other)
Responsible Party: Sponsor
Other Study IDs: CM0118-PLI-3
Record Dates: First submitted 2018-06-26; First posted 2018-07-30 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2019-12

CONDITIONS: Coronary Stenosis; Acute Coronary Syndrome; Acute Myocardial Infarction; Atheromatous Plaques; Atheroscleroses, Coronary; Non-ST Elevation Myocardial Infarction (nSTEMI)
Keywords: coronary artery disease; myocardial infarction; cardiac imaging techniques; major adverse cardiovascular events; vulnerable coronary plaques; serum biomarkers; coronary shear stress
MeSH Terms: conditions — Coronary Stenosis; Acute Coronary Syndrome; Plaque, Atherosclerotic; Coronary Artery Disease; Non-ST Elevated Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood sample collection during the acute coronary event for evaluation of serum levels of hsCRP, IL-6, matrixmetalloproteases MMP9, Adhesion molecules (VCAM, ICAM), hs-cTnI, NTproBNP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VP-SG 01: Study subjects that present MACE at the 36 months follow-up
  Interventions: Diagnostic Test: Cardiac imaging tests; Diagnostic Test: Venous blood sample collection
- VP-SG 02: Study subjects that do not present MACE at the 36 months follow-up
  Interventions: Diagnostic Test: Cardiac imaging tests; Diagnostic Test: Venous blood sample collection

INTERVENTIONS:
Diagnostic Test: Cardiac imaging tests — * 2D transthoracic echocardiography
  * 128-multislice CT coronary angiography with the evaluation of: epicardial fat volume, plaque burden, total and local calcium score, markers for lesion severity; morphological plaque characteristics; plaque components evaluated via volumetric and planimetric units; markers of plaque vulnerability (necrotic core, low attenuation plaque, spotty calcification, napkin ring sign, positive remodeling).
  * Shear stress evaluation via computational fluid dynamics.
  * Intracoronary imaging techniques: IVUS and OCT.
Diagnostic Test: Venous blood sample collection — Venous blood sample collection during the acute coronary event for evaluation of serum levels of hsCRP, IL-6, matrixmetalloproteases MMP9, Adhesion molecules (VCAM, ICAM), alfa tumour necrosis factor, hs-cTnI, NTproBNP

SUMMARY:
• The aim of the VIP study is to investigate the impact of vulnerability markers (inflammatory serum biomarkers for systemic vulnerability, coronary shear stress and vulnerability mapping for pancoronary vulnerability, and imaging-based plaque features for systemic vulnerability) on the rate of major adverse cardiovascular events caused by progression of the non-culprit lesion in patients with acute ST or non-ST segment elevation myocardial infarction who undergo revascularization of the culprit lesion during the acute event. Furthermore, the study will evaluate the rate of progression of non-culprit lesions towards a higher degree of vulnerability, based on coronary computed tomography angiographic assessment at 1 year after enrollment.

DETAILED DESCRIPTION:
The project is a prospective, cohort, mono-centric study which will be carried out in the Center of Advanced Research in Multimodal Cardiac Imaging Cardiomed.

The project will include 100 subjects who present ST and non-ST segment elevation myocardial infarction at 30 days prior to study enrollment, who underwent emergency revascularization of the culprit lesion. Samples for systemic serum biomarkers for myocardial injury, myocardial strain and enhanced systemic inflammation will be collected at the moment of the acute event. All patients will undergo coronary CT angiography, cardiac perfusion CT and intracoronary imaging procedures (Intravascular ultrasound - IVUS; Optical Coherence Tomography - OCT) at the moment of enrollment in the study, for complex assessment of non-culprit coronary lesions. The endothelial coronary shear stress will be calculated with imaging post-processing techniques on the CT data acquired at baseline, by using computational fluid dynamics.

The study will be conducted over a period of 3 years, in which patients will be examined at baseline, and during several follow-up visits. At the one-year follow-up, the study subjects will undergo CT coronary angiography for re-evaluation of the non-culprit lesions, in the prospects of analyzing the rate of plaque progression towards a higher degree of vulnerability. At the end of the 3-year period, patients will be assessed about the occurrence of major adverse cardiovascular events and the rate or revascularization for non-culprit lesions.

Study objectives:

Primary: to investigate the association between systemic, pancoronary and local vulnerability features of coronary plaques and the risk for major adverse cardiac events - MACE (all-cause mortality, cardiovascular death, myocardial infarction, repeated revascularization, repeated hospitalizations for cardiovascular related incidents, cerebrovascular events) during a 3-year follow-up.

Secondary: to assess the rate of progression for the non-culprit lesions towards a higher degree of vulnerability, as evaluated via coronary CT angiography at 1 year after enrollment, in relation to systemic, pancoronary and local vulnerability features at baseline.

To identify the type of vulnerability (systemic, pancoronary or local) with the highest impact on plaque progression and future MACE

Study Timeline:

Baseline (day 0)

* Obtain and document consent from participant on study consent form.
* Verify inclusion/exclusion criteria.
* Obtain demographic information, medical history, medication history, alcohol and tobacco use history.
* Record results of physical examinations and 12-lead ECG.
* Collect blood specimens.
* Imaging procedures: transthoracic 2-D echocardiography, 128-multisclice CT angiography, cardiac perfusion CT, IVUS, OCT

Visit 1 (month 1)

* Record results of physical examinations, 12-lead ECG and medical history.
* Imaging procedures: transthoracic 2-D echocardiography

Visit 2 (month 3)

• Telephone follow-up

Visit 3 (month 6)

* Record results of physical examinations, 12-lead ECG and medical history.
* Imaging procedures: transthoracic 2-D echocardiography

Visit 4 (month 12)

* Record results of physical examinations, 12-lead ECG and medical history.
* Imaging procedures: transthoracic 2-D echocardiography, 128-multislice CT coronary angiography for evaluation of non-culprit lesion
* End-point evaluation

Visit 5 (month 15)

• Telephone follow-up

Visit 6 (month 18)

• Telephone follow-up

Visit 7 (month 24)

* Record results of physical examinations, 12-lead ECG and medical history.
* Imaging procedures: transthoracic 2-D echocardiography.
* End-point evaluation

Visit 8 (month 30)

• Telephone follow-up

Final study visit (month 36)

* Record results of physical examinations, 12-lead ECG and medical history.
* Imaging procedures: transthoracic 2-D echocardiography
* End-point evaluation.

Study procedures:

* Clinical examination, medical history
* 12-lead ECG
* 2D transthoracic echocardiography with measurement of: cardiac diameters, volumes, valvular function and regurgitation, pressure gradients, pericardial fat thickness, pericardial effusion, left ventricular global and regional function and ejection fraction.
* 128-multislice CT coronary angiography with the evaluation of: epicardial fat volume, plaque burden, total and local calcium score, markers for lesion severity (degree of stenosis, lesion length, lumen area and diameter, minimum and maximum plaque thickness); morphological plaque characteristics (plaque related volumes, plaque burden, vascular indexes - remodeling and eccentricity index); plaque components evaluated via volumetric and planimetric units (necrotic core, fibrofatty tissue, fibrotic tissue, dense calcium); markers of plaque vulnerability (necrotic core, low attenuation plaque, spotty calcification, napkin ring sign, positive remodeling).
* Shear stress evaluation of CT acquired images and computational fluid dynamics
* Intracoronary imaging techniques: IVUS and OCT with evaluation of plaque characteristics.
* Venous blood sample collection during the acute coronary event for evaluation of serum levels of hsCRP, IL-6, matrixmetalloproteases MMP9, Adhesion molecules (VCAM, ICAM), alfa tumour necrosis factor, hs-cTnI, NTproBNP

Data collection: In a dedicated database that includes all patient information, demographics, medical history, medication, therapeutic procedures, information derived from imaging techniques (echocardiography, CT angiography, CT imaging post-processing and shear stress evaluation).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old that have signed the written informed consent;
* Patients with ST and non-ST segment elevation myocardial infarction (as stated in the Third Universal Definition of Myocardial Infarction) at 30 days prior to randomization;

Exclusion Criteria:

* unwillingness or incapacity to provide informed consent (and if consent of legal guardian or family is not available);
* acute myocardial infarction at the moment of randomization (as these patients are referred to the hospital for emergency invasive coronary angiography and revascularization)
* conditions that present an estimated life expectancy of under 5 years;
* acute renal failure or terminal stage chronic kidney disease;
* pregnancy or lactation and women of reproductive age who are not using any contraceptive method;
* allergy and history of allergic reactions to iodine contrast media;
* active malignancy or malignancy within the last 1 year prior to enrollment;
* patients who, in the opinion of the investigators are not compliant and will not present for study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with present ST and non-ST segment elevation myocardial infarction at 30 days prior to study enrollment, who underwent emergency revascularization of the culprit lesion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
MACE rate - Major adverse cardiovascular events | 36 months
  Acute coronary syndromes (unstable angina, ST and non-ST elevation myocardial infarction), emergency revascularization of non-culprit lesions, repeated hospitalizations for cardiovascular reasons, acute cerebrovascular event.

SECONDARY OUTCOMES:
Severity progression of non-culprit coronary lesions | 12 months
  Reevaluation of the non-culprit lesions via 128-multislice CT coronary angiography with analysis of the degree of stenosis caused by the non-culprit lesion.
Progression rate of CT markers for coronary plaque vulnerability | 12 months
  Reevaluation of the non-culprit lesions via 128-multislice CT coronary angiography with analysis of the number of CT markers for coronary plaque vulnerability (low attenuation plaque, spotty calcification, napkin ring sign, positive remodeling).

CONTACTS AND LOCATIONS:
Overall Officials: Theodora Benedek, Professor, Study Director — Cardio Med Medical Center
Locations (1):
- Cardio Med, Târgu Mureş, Mureș County, Romania

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available for interested parties.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The IPD sharing frame is starting 6 months after publication.